CLINICAL TRIAL: NCT00412269
Title: Healthy Transitions: Menopause Effect on Obesity, Energy Balance, and Insulin
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Donna H. Ryan, MD, Professor, Adjunct, Pennington Biomedical Research Center
Other Study IDs: PBRC 97022
Record Dates: First submitted 2006-12-14; First posted 2006-12-18 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Menopause
Keywords: Insulin Sensitivity; Total abdominal fat; Visceral abdominal fat; Reproductive Hormones; Menopause; Diabetes; Fat Distribution; Sex Hormones
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine the effect of menopause on obesity, energy balance, and insulin in postmenopausal, obese women.

DETAILED DESCRIPTION:
The effect of menopause on body composition and cardiovascular risk in healthy caucasian women has been the subject of much study. In contrast, there are few data available on menopause in African-American women. Since menopause is associated with potentially preventable health risks in women, this proposal is aimed at characterizing the perimenopausal period in terms of body fat, energy balance, and insulin action in both caucasian and African-American women.

The study will address 4 general hypotheses:

* Menopause increases both total and visceral abdominal fat
* Changes in body composition and body weight at menopause are mediated, at least in part by changes in 24-hour energy expenditure and/or food intake
* Menopause results in decreased insulin sensitivity that may predispose certain women to develop diabetes later in life
* African-American women may respond to the shifts in reproductive hormones at menopause differently than caucasian women.

ELIGIBILITY:
Inclusion Criteria:

* Age 47-52 yr, at time of enrollment
* Body Mass Index 25-40
* Normal oral glucose tolerance test by National Diabetes Data Group criteria
* Premenopausal, defined by FSH levels <30mIU/ml and at least 5 menstrual periods in the last 6 months
* Able to confirm ethnic heritage of past 2 generations in family

Exclusion Criteria:

* hypertension or hypercholesterolemia requiring medication
* regular use of medications that influence glucose tolerance
* use of oral contraceptives within the past 6 months
* history of myocardial infarction or significant coronary vascular disease or stroke
* history of endocrine, kidney, or liver disease or malignancy
* any psychopathology, including eating disorders, substance abuse, and major depression
* unable to complete longitudinal study commitment, including anticipating moving out of the area within the next 5 years.

Ages: 47 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pennington Biomedical Research Center is located in Baton Rouge, Louisiana, adjacent to the medical services district of the Regional Medical Center. The city of Baton Rouge is the home of state government, the 27,000-student Louisiana State University, the 9,000-student Southern University and a large petrochemical industry. Lacking the traditional active urban "downtown", the region is characterized by the suburban pattern of single family subdivisions and small apartment complexes. The population within a 7 parish (i.e. county) area is 635,202. The population of East Baton Rouge Parish is 380,105 with an ethnic distribution of 62% Caucasian, 35% African-American, 1% Asian, and <1% Native American and Hispanic. There are 34,885 people over age 65 and 251,586 between ages 16-65 yr.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 1998-02; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Smith, M. D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Lovejoy JC, Champagne CM, de Jonge L, Xie H, Smith SR. Increased visceral fat and decreased energy expenditure during the menopausal transition. Int J Obes (Lond). 2008 Jun;32(6):949-58. doi: 10.1038/ijo.2008.25. Epub 2008 Mar 11. PMID 18332882